CLINICAL TRIAL: NCT04983394
Title: Effect of Motion-Controlled Video Games-Based Virtual Reality Exercise On Pain, Fatigue, Mood, Functional Capacity, And Quality of Life in Patients With Post-Covid-19 Condition: A Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality Exercises on Patients With Post-COVID-19 Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, MUSA POLAT, Principal Investigator, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SivasCumhuriyetUniversity
Record Dates: First submitted 2021-07-28; First posted 2021-07-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Realty (Experimental): Virtual reality exercises were implemented semi-immersively in the Kinect Sports Rivals program via the Microsoft Xbox One Kinect game console and Kinect V2 infrared camera. Participants were positioned 2 meters away from a 55-inch LCD screen in a well-lit room. Motion-controlled video games, including tennis, bowling, soccer, target shooting, climbing, and jet ski racing, were played against a virtual opponent, starting at a basic difficulty level and increasing in difficulty based on the participant's ability to defeat their opponent. Game transitions and difficulty adjustments were provided by the physical therapist. Participants performed plyometric movements such as jumping and shooting, as well as limb and spine movements, to direct the avatar and ensured the coordination of their movements.
  Interventions: Other: Virtual Realty Exercises
- Conventional (Active Comparator): Flexibility exercises were performed during the warm-up and cool-down periods of aerobic exercise for 3-5 minutes, consisting of static and dynamic upper and lower extremity stretching exercises in standing and sitting positions. Neuromuscular exercises were performed on the Bosu ball and balance board with eyes open and closed, using one or both feet.
  Aerobic exercise using a bicycle ergometer was performed for 20-30 minutes, depending on patient tolerance, starting at 60% of the age-determined maximum heart rate and increasing by 5% every 2 weeks (75% in the last 2 weeks).
  Strengthening exercises were performed for 10-15 minutes using dumbbells or sandbags targeting the large muscles of the upper and lower extremities. Initially, one set of strengthening exercises was performed with 8 repetitions targeting 6 different muscles at 50% of 1 RM intensity. Depending on patient tolerance, the exercise intensity was increased weekly to 70%, the number of muscles worked to 10, the number o
  Interventions: Other: conventional exercises

INTERVENTIONS:
Other: Virtual Realty Exercises — motion-controlled video game
  Arms: Virtual Realty
Other: conventional exercises — aerobic, strength, stretching, and neuromuscular exercises
  Arms: Conventional

SUMMARY:
This study aims to investigate (I) the effectiveness of motion-controlled video game-based VR exercises on pain, fatigue, functional capacity, mood, and quality of life in patients with PCC, and (II) to determine whether they are superior to conventional exercise.

DETAILED DESCRIPTION:
79 individuals aged 18-65 years who were diagnosed with COVID-19 with a PCR test result in an oropharyngeal or nasopharyngeal swab sample taken more than 90 days ago and who had PCC symptoms for at least eight weeks were included. Patients with PCC who had been hospitalized, had signs of pneumonia or organ failure, had suffered an acute myocardial infarction or orthopedic surgery within the last 2 years, had cardiovascular system diseases such as uncontrolled hypertension, arrhythmia, or cardiac insufficiency, had known chronic respiratory system diseases, those with conditions causing widespread pain such as fibromyalgia syndrome, those with primary any neurological system diseases, or those unable to mobilize for any reason were excluded from the study.

The same physiatrist systematically evaluated the sociodemographic data, medical history including the time elapsed since the diagnosis of COVID-19, the duration of PCC symptoms, and outcome measures (fatigue level, pain intensity, general health status, emotional state, functional capacity) through face-to-face interviews at the hospital, and recorded in a standardized form.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with COVID-19 by polymerase chain reaction from an oropharyngeal or nasopharyngeal swab sample more than 90 days ago, and who had PCC symptoms for at least eight weeks

Exclusion Criteria:

* have been hospitalized due to COVID-19,
* have developed pneumonia or organ failure findings.
* have had an acute myocardial infarction in the last 2 years,
* have cardiovascular system disease such as uncontrolled hypertension, arrhythmia, aneurysm, cardiac failure,
* have undergone fracture or orthopedic surgery in the last 2 years,
* have a known chronic respiratory system disease,
* have widespread pain such as fibromyalgia syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
visual Analogue Scale | 8th week

SECONDARY OUTCOMES:
hospital anxiety and depression scale-Depression | 0th and 8th week
hospital anxiety and depression scale-Anxiety | 0th and 8th week
Fatigue severity scale | 0th and 8th week
Short Form-12 | 0th and 8th week
6 minutes walking test | 0th and 8th week

CONTACTS AND LOCATIONS:
Overall Officials: Musa Polat, Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The plan will be shared by the corresponding author at the submission stage if requested.